CLINICAL TRIAL: NCT00822432
Title: Urinary Ratio of the Coproporphyrins Isomers I and III and Its Relationships With Methotrexate Elimination in Patients With a Lymphoid Malignancy
Brief Title: Coproporphyrine Isomers and Methotrexate Elimination
Acronym: COMETH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P061005
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2009-01

CONDITIONS: Central Nervous System Neoplasms; Lymphoma, Large B-Cell, Diffuse; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma
Keywords: biomarkers; ABC transporters; MRP2; MTX pharmacokinetics
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma, Large B-Cell, Diffuse; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1

SUMMARY:
High dose methotrexate (MTX) is responsible of severe toxicity in patients in whom elimination from plasma is delayed. Factors responsible for MTX accumulation are partly known but some patients still experience toxicity despite adequate measures being taken. Our hypothesis is that renal tubular secretion may be impaired in these patients. This study aims at evaluating the performance of the UCP ratio (urinary ratio of coproporphyrins), a putative biomarker of tubular secretion, in predicting delayed MTX elimination.

DETAILED DESCRIPTION:
MTX is a substrate of MRP2, a renal tubular transporter encoded by the ABCC2 gene. It has been shown that single nucleotide polymorphisms (SNPs) on the ABCC2 gene are associated with impairment of MTX elimination. Mutations on the ABCC2 gene are also responsible for the Dubin-Johnson syndrome, characterised by the absence of a functional MRP2 protein. Apart from hyperbilirubinaemia, the main biological perturbation observed in this disease is a typical increase of the urinary ratio of coproporphyrins I (I+ III) (UCP ratio). Our hypothesis is that the UCP ratio could be used as a biomarker of MRP2's activity, thus predicting MTX elimination. One hundred patients treated with high dose MTX will be recruited in this prospective study. Their UCP ratio will be measured before and after MTX administration and correlated with MTX clearance. A genetic analysis will be conducted to study the five more frequents SNPs of ABCC2 in each patient.

ELIGIBILITY:
Inclusion criteria :

* Patients receiving HDMTX (≥1g/m2) for a primitive cerebral lymphoma, a large cell lymphoma, a lymphoblastic lymphoma, a Burkitt's lymphoma or an acute lymphoblastic leukaemia,
* over 18 years old,
* Signed informed consent.
* Affiliated to a medical assurance.
* Able to respect the protocol.
* Effective contraception for women.

Exclusion criteria :

* renal failure,
* liver failure,
* hepatic cytolysis,
* chronic respiratory deficiency,
* pregnancy,
* breast-feeding,
* Concomitant medication: phenytoin, probenecid, trimethoprim, phenylbutazone, salicylates, non steroid anti-inflammatory, yellow fever vaccine.
* Patient included in another study in the four weeks preceding his inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients aged more than 18 y, hospitalized in the neurology or in the haematology department at PSP hospital of Paris or in the haematology department at CHU of Tours
  * Who should receive high-dose methotrexate (> 1 g/m2) for one of the following conditions : Central Nervous System Neoplasms; Lymphoma, Large B-Cell, Diffuse; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma or Burkitt lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2007-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
MTX concentrations | at the end of MTX infusion and every 24-hours until concentrations reach 0,2µM.

SECONDARY OUTCOMES:
The UCP I/(I+III) ratio | before and at the end of MTX infusion and at the end of hospitalisation.
Five polymorphisms of the ABCC2 gene (-24C/T, 1249G/A, 3563T/A, 4544G/A) | during the study
Blood cells count . | before MTX infusion and at the end of hospitalisation
Renal function | before MTX infusion and at the end of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Le Guellec, PharmD, PhD, Principal Investigator — CHRU of Tours
Locations (2):
- France (2):
  - Pitié-Salpêtrière Hospital, Paris
  - University Hospital Centre of Tours, Tours

REFERENCES:
- [Derived] Benz-de Bretagne I, Zahr N, Le Gouge A, Hulot JS, Houillier C, Hoang-Xuan K, Gyan E, Lissandre S, Choquet S, Le Guellec C. Urinary coproporphyrin I/(I + III) ratio as a surrogate for MRP2 or other transporter activities involved in methotrexate clearance. Br J Clin Pharmacol. 2014 Aug;78(2):329-42. doi: 10.1111/bcp.12326. PMID 24433481